CLINICAL TRIAL: NCT01720485
Title: A Double-blind,Double Dummy, Randomized, Multicenter Parallel-group Study on Efficacy of Desloratadine and Prednisolone Association Compared to Dexchlorpheniramine and Betamethasone Association in Adults With Moderate - Severe Persistent Allergic Rhinitis
Brief Title: Comparison of Desloratadine Associated With Prednisolone (Tablet)Versus Dexchlorpheniramine Associated With Betamethasone (Tablet) for Adult Persistent Allergic Rhinitis Treatment
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DPCEMS0812
Record Dates: First submitted 2012-10-31; First posted 2012-11-02 (Estimated); Last update posted 2013-09-25 (Estimated); Status verified 2013-09

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — desloratadine; Prednisolone; dexchlorpheniramine; Betamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Desloratadine + Prednisolone (Experimental): The patients will take 2 tablets three times a day, as follows:
  Morning: 1 tablet of the test medication(Desloratadine 5 mg + Prednisolone 20 mg) + 1 tablet of placebo control medication.
  Afternoon: 1 tablet of placebo test medication + 1 tablet of placebo control medication.
  Night: 1 tablet of placebo test medication + 1 tablet of placebo control medication.
  Interventions: Drug: Desloratadine + Prednisolone
- Dexchlorpheniramine + Betamethasone (Active Comparator): The patients will take 2 tablets three times a day, as follows:
  Morning: 1 tablet of the control medication(Dexchlorpheniramine 2mg + Betamethasone 0.25mg) + 1 tablet of placebo test medication.
  Afternoon: 1 tablet of the control medication(Dexchlorpheniramine 2mg + Betamethasone 0.25mg) + 1 tablet of placebo test medication.
  Night: 1 tablet of the control medication(Dexchlorpheniramine 2mg + Betamethasone 0.25mg) + 1 tablet of placebo test medication.
  Interventions: Drug: Dexchlorpheniramine + Betamethasone

INTERVENTIONS:
Drug: Desloratadine + Prednisolone — 1 tablet 3 times a day
  Arms: Desloratadine + Prednisolone
Drug: Dexchlorpheniramine + Betamethasone — 1 tablet 3 times a day
  Arms: Dexchlorpheniramine + Betamethasone

SUMMARY:
The purpose of this study is to evaluate the non-inferiority clinical efficacy of two different drug associations in the treatment of Moderate - Severe Persistent Allergic Rhinitis in Adults.

ELIGIBILITY:
Inclusion Criteria:

* Signed Consent of the patient;
* Clinical diagnosis of moderate - severe persistent allergic rhinitis according to ARIA classification(Allergic Rhinitis and Its Impact on Asthma);
* Adults aged ≥ 18 years old;
* Evidence of sensitization to aeroallergens in examination (immediate skin tests or serum specific IgE) in the 12 months prior to inclusion.

Exclusion Criteria:

* Decongestants dependent patients or patients receiving allergen specific immunotherapy;
* Patients who were in use of oral antihistamines or decongestants in the past 15 days;
* Patients who were treated with systemic corticosteroids in the last month;
* Patients on treatment with monoamine oxidase inhibitors (MAOIs);
* Patients with history of hypersensitivity to any of the formula compounds;
* Patients with any clinically significant disease that in the investigator opinion can not participate in the study
* Patients who have uncontrolled asthma, chronic sinusitis, drug related rhinitis and nasal anatomic abnormalities.
* Participation in clinical trial in 30 days prior to study entry;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2013-10; Primary Completion 2013-12 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy of treatment in persistent allergic rhinitis based on nasal symptoms score | 7 days
  The mean variability of nasal symptoms score observed between visit 1 and visit 2 will be used as the primary endpoint of clinical efficacy.

SECONDARY OUTCOMES:
Safety will be evaluated by the adverse events occurrences | 7 days
  Adverse events will be collected and followed in order to evaluate safety and tolerability

CONTACTS AND LOCATIONS:
Locations (1):
- IMA - Instituto de Pesquisa Clínica e Medicina Avançada, São Paulo, Brazil